CLINICAL TRIAL: NCT03509311
Title: Investigation of Physical Activity Level, Cardiorespiratory Fitness and Quality of Life in Patients With Asthma
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof., Gazi University
Other Study IDs: Gazi University 11
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Asthma; Physical Activity
Keywords: Asthma; Physical activity; Cardiorespiratory fitness; Quality of life
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma Group: That group consists from patients who had diagnosed as asthma by doctors from Chest Diseases Department of Gazi University Hospital.
  Physical activity level assesment, maximal and submaximal exercise capacity assesment, respiratory function assesment, respiratory muscle strength assesment, respiratory muscle endurance assesment, peripheral muscle strength assesment, quality of life assesment about disease specific, respiratory, sleep and cough associated, fatigue severity assesment, depression and anxiety level assesment and asthma management knowledge assesment apply to this group.
- Healthy Group: That group consists from participants who do not have any diagnosed disease. Physical activity level assesment, maximal and submaximal exercise capacity assesment, respiratory function assesment, respiratory muscle strength assesment, respiratory muscle endurance assesment, peripheral muscle strength assesment, quality of life assesment about disease specific, respiratory, sleep and cough associated, fatigue severity assesment and depression and anxiety level assesment apply to this group.

SUMMARY:
The primary aim of the study is to evaluate the physical activity level in patients with asthma. The secondary aims of the study are assesment of maximal and functional exercise capacity, respiratory functions, respiratory muscle strength and endurance, peripheral muscle strength, depression and anxiety levels, disease specific and respiratory quality of life, sleep and coughing associated quality of life, asthma self-management knowledge level and fatigue severity in patients with asthma.

DETAILED DESCRIPTION:
Asthma is an obstructive pulmonary disease and thus it affects respiratory functions. Dyspnea, fatigue and bronchial hyperreactivity symptoms are commonly seen on patients with asthma. It is known that physical activity level of asthmatic patients is reduced. Few researches have investigated asthmatic patients' physical activity level and these researches mainly focused on self reported physical activity level. How differing maximal and submaximal exercise capacity of asthmatic patients is not well known. Because previous researches compared only different severity levels of the disease. It is reported that peripheral muscle strength of asthmatic patients is lower than healthy individuals' peripheral muscle strength. But evidences about this subject are insufficient. Asthmatic patients' respiratory muscle strength is lower than healthy individuals' respiratory muscle strength. But it is not clear if endurance is lower as respiratory muscle strength too, or not. It is reported that quality of life of asthmatic patients is worst than healthy individuals'. According to the sample size analysis 36 patients and 36 healthy individuals with similar demographic characteristics will be included the study. Patients and healthy individuals will be selected according to predetermined inclusion and exclusion criteria. The assessments will be completed in two days. Maximal exercise capacity will be assessed using cardiopulmonary exercise testing (CPET), functional exercise capacity using six minute stepper test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, depression using Beck Depression Inventory (Turkish version), anxiety using Beck Anxiety Inventory (Turkish version), disease specific quality of life using Asthma Quality of Life Questionnaire (Turkish version) and St. George Respiratory Questionnaire (Turkish version), cough related quality of life using Leicester Cough Questionnaire (Turkish version), sleep related quality of life using Pittsburgh Sleep Quality Index (Turkish version), asthma control level using Asthma Control Test (Turkish version), disease management knowledge level using Asthma Self-Management Questionnaire (Turkish version).

ELIGIBILITY:
Inclusion criteria for asthma group: Patients who are;

* Between 18-65 years
* Diagnosed with asthma
* Receiving standard medical treatment
* Asthma Control Test score ≥ 20 point
* No smoker or ex-smoker (if ex-smoker, smoke exposure below 10 packyears)
* Willing to participate in the study

Exclusion criteria for asthma group: Patients who are;

* Have cooperation difficulty
* Have pulmonary disease (except asthma for asthma group)
* Have any cardiac, neurological or orthopedic disease that affects functional capacity
* Have pneumonia or acute infection (at last one month)
* Have been used oral corticosteroids at last one year
* Have any psychiatric diseases
* Refusing to participate
* Received or are receiving non-standard medical treatment will be excluded from study.

Inclusion criteria for healthy group: Participants who are;

* Between 18-65 years without any diagnosed disease
* No smoker or ex-smoker (if ex-smoker, smoke exposure below 10 packyears)
* Willing to participate in the study will be included in healthy group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For Asthma Group:
  Thirty six patients with asthma will be included in this group
  For Healthy Group:
  Thirty six healthy volunteer will be included in this group.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | First Day
  Multi sensor activity monitor

SECONDARY OUTCOMES:
Pulmonary Functions | First Day
  Spirometry
Respiratory Muscle Strength | First Day
  Mouth pressure meter
Respiratory Muscle Endurance | First day
  Incremental threshold loading test
Peripheral Muscle Strength | First Day
  Hand held dynamometer
Disease Spesific Quality of Life | First Day
  Asthma Quality of Life Questionnaire (Turkish version) (disease specific) - Asthma Quality of Life Questionnaire (AQLQ) is a self-reported questionnaire. AQLQ evaluates disease spesific quality of life. This questionnaire includes 32 items and 4 subcategories [Symptoms (11 items), Activity Limitation (12 items, 5 of which are individualized), Emotional Function (5 items), and Environmental Exposure (4 items)] . Score range for each item from 1 to 7 point (7-point Likert scale). Higher scores show fine quality of life.
Fatigue Severity | First Day
  Fatigue Severity Scale (Turkish version) - Fatigue Severity Scale (FSS) is a self-reported questionnaire. FSS evaluates patient's fatigue severity. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Asthma Self-Management Knowledge | First Day
  Asthma Self-Management Knowledge Questionnaire (Turkish version) - Asthma Self-Management Knowledge Questionnaire (AKQ) is a self-reported questionnaire. AKQ evaluates patients' knowledge level about disease management. This questionnaire includes 24 items about general asthma knowledge, asthma medications, asthma exacerbations, and environmental triggers, with responses of "true" or "false". This questionnaire scored as counting correct answers. As scoring this questionnaire more correct answer indicates higher knowledge about self-management of disease.
Functional Exercise Capacity | First Day
  Six minute stepper test
Maximal Exercise Capacity | Second Day
  Cardiopulmonary exercise testing (Oxygen consumption measurement during test)
Anxiety | Second Day
  Beck Anxiety Inventory (Turkish version) - Beck Anxiety Inventory (BAI) is a self-reported questionnaire. BAI evaluates patients' anxiety level. This questionnaire includes 21 items. Each item scores from 0 to 3 point (higher scores shows more severe anxiety). The BAI scores are classified as minimal anxiety (0 to 7), mild anxiety (8 to 15), moderate anxiety (16 to 25), and severe anxiety (30 to 63).
Depression | Second day
  Beck Depression Inventory (Turkish version) - Beck Depression Inventory (BDI) is a self-reported questionnaire. BDI evaluates patients' depression level. This questionnaire includes 21 items. Each item scores from 0 to 3 point (higher scores shows patient ). The BAI scores are classified as "depression" over 17 points.
Respiratory Associated Quality of Life (respiratory) | Second day
  St. George Respiratory Questionnaire (Turkish version) (respiratory) - St. George Respiratory Questionnaire (SGRQ) is a self-reported questionnaire. SGRQ evaluates patients' respiratory disease associated quality of life. This questionnaire includes 2 part (part one is about symptoms (one subsection) and part two is about activity (seven subsection)) and 50 items. Some items scored as Likert scale and others scored as dichotomous (true/false).
Sleep Quality | Second day
  Pittsburgh Sleep Quality Index (Turkish version) - Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire. PSQI evaluates patients' sleep quality. The scale includes 24 questions overall, with 19 questions answered by the person him/ herself and the remaining 5 answered by his/her bed partner or roommate. The first 19 self-answered questions evaluate 7 subscales, subjective sleep quality, sleep latency, duration of sleep, routine sleep activity, sleep disorders, the use of drugs for sleeping, and daytime dysfunction. Each item in the scale is scored between 0 and 3 (no difficulty to severe difficulty). The sum of the 7 subscale scores gives the overall PSQI score. Lower scores show better sleep quality.
Cough Related Quality of Life | Second day
  Leicester Cough Questionnaire (Turkish version) - Leicester Cough Questionnaire (LCQ) is a self-reported questionnaire. LCQ evaluates patients' quality of life about cough symptom. This questionnaire includes 19 items and score range for each item from 1 to 7 point (7-point Likert scale). Higher scores show better quality of life about cough symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Ozdemir, PT, Study Chair — Gazi University; Meral Bosnak Guclu, Assoc. Prof, Study Director — Gazi University; Hanim Eda Goktas, PhD, Principal Investigator — Gazi University; I. Kivilcim Oguzulgen, MD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bruno A, Uasuf CG, Insalaco G, Barazzoni R, Ballacchino A, Gjomarkaj M, Pace E. Nutritional status and physical inactivity in moderated asthmatics: A pilot study. Medicine (Baltimore). 2016 Aug;95(31):e4485. doi: 10.1097/MD.0000000000004485. PMID 27495092
- [Background] Shei RJ, Paris HL, Wilhite DP, Chapman RF, Mickleborough TD. The role of inspiratory muscle training in the management of asthma and exercise-induced bronchoconstriction. Phys Sportsmed. 2016 Nov;44(4):327-334. doi: 10.1080/00913847.2016.1176546. Epub 2016 Apr 26. PMID 27094568
- [Background] Ramos E, de Oliveira LV, Silva AB, Costa IP, Correa JC, Costa D, Alves VL, Donner CF, Stirbulov R, Arena R, Sampaio LM. Peripheral muscle strength and functional capacity in patients with moderate to severe asthma. Multidiscip Respir Med. 2015 Jan 21;10(1):3. doi: 10.1186/2049-6958-10-3. eCollection 2015. PMID 25973197
- [Background] Vargas Becerra MH. [Physiopathology of asthma]. Rev Alerg Mex. 2009;56 Suppl 1:S24-8. Spanish. PMID 20873050
- [Background] Fitting JW. [Fatigue of the respiratory muscles]. Schweiz Med Wochenschr. 1992 Feb 29;122(9):302-6. French. PMID 1546280
- [Background] Cluley S, Cochrane GM. Psychological disorder in asthma is associated with poor control and poor adherence to inhaled steroids. Respir Med. 2001 Jan;95(1):37-9. doi: 10.1053/rmed.2000.0968. PMID 11207015
- [Background] Stucky BD, Sherbourne CD, Edelen MO, Eberhart NK. Understanding asthma-specific quality of life: moving beyond asthma symptoms and severity. Eur Respir J. 2015 Sep;46(3):680-7. doi: 10.1183/09031936.00225014. Epub 2015 Apr 16. PMID 25882804